CLINICAL TRIAL: NCT01611311
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Rising Doses of BI 409306 Film-coated Tablets Given Orally q.d. for 14 Days in Young and Elderly Healthy Male/Female Volunteers (Randomized, Double-blind, Placebo Controlled Within Dose Groups Phase I Study)
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Rising Doses of BI 409306
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1289.17; 2012-000052-34 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-05-22; First posted 2012-06-04 (Estimated); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — BI 409306

ARMS (6):
- Placebo (Young subjects) (Placebo Comparator): Young healthy subjects received placebo matching film-coated tablets of BI 409306 orally after an overnight fast once daily for 14 days
  Interventions: Drug: Placebo
- BI 409306 - 25 milligram (mg) (Young subjects) (Experimental): Young healthy subjects received 25 mg of BI 409306 film-coated tablets orally after an overnight fast once daily for 14 days
  Interventions: Drug: BI 409306
- BI 409306 - 50 milligram (mg) (Young subjects) (Experimental): Young healthy subjects received 50 mg of BI 409306 film-coated tablets orally after an overnight fast once daily for 14 days
  Interventions: Drug: BI 409306
- Placebo (Elderly subjects) (Placebo Comparator): Elderly healthy subjects received placebo matching film-coated tablets of BI 409306 orally after an overnight fast once daily for 14 days
  Interventions: Drug: Placebo
- BI 409306 - 25 milligram (mg) (Elderly subjects) (Experimental): Elderly healthy subjects received 25 mg of BI 409306 film-coated tablets orally after an overnight fast once daily for 14 days
  Interventions: Drug: BI 409306
- BI 409306 - 50 milligram (mg) (Elderly subjects) (Experimental): Elderly healthy subjects received 50 mg of BI 409306 film-coated tablets orally after an overnight fast once daily for 14 days
  Interventions: Drug: BI 409306

INTERVENTIONS:
Drug: BI 409306 — Film-coated tablet
  Arms: BI 409306 - 25 milligram (mg) (Elderly subjects); BI 409306 - 25 milligram (mg) (Young subjects); BI 409306 - 50 milligram (mg) (Elderly subjects); BI 409306 - 50 milligram (mg) (Young subjects)
Drug: Placebo — Elderly healthy subjects received 50 mg of BI 409306 film-coated tablets orally after an overnight fast once daily for 14 days
  Arms: Placebo (Elderly subjects); Placebo (Young subjects)

SUMMARY:
The primary objective of the current study is to investigate the safety and tolerability of BI 409306 in healthy young and elderly male and female volunteers following oral administration of repeated rising doses, given once daily over 14 days to young healthy genotyped and elderly healthy male/female volunteers.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male/female subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2012-08-01 (Actual); Study Completion 2012-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1289.17.1 Boehringer Ingelheim Investigational Site, Neuss, Germany

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Safety, tolerability, pharmacokinetics, and pharmacodynamics of multiple rising doses of BI 409306 film-coated tablets given orally once daily (q.d.) for 14 days in young and elderly healthy male/female volunteers (randomized, double-blind, placebo controlled within dose groups Phase I study).All young subjects were Poor Metabolizer for CYP2C19
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended a specialist sites which ensured that they met all strictly implemented inclusion/exclusion criteria. Subjects were not to be entered to trial if any one of the specific entry criteria was violated.
Period: Overall Study
Arm/Group | Placebo (Young Subjects) | BI 409306 - 25 Milligram (mg) (Young Subjects) | BI 409306 - 50 Milligram (mg) (Young Subjects) | Placebo (Elderly Subjects) | BI 409306 - 25 Milligram (mg) (Elderly Subjects) | BI 409306 - 50 Milligram (mg) (Elderly Subjects)
Started | 4 | 6 | 6 | 6 | 9 | 9
Completed | 4 | 6 | 6 | 6 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The treated set (TS) included all subjects who were randomised and documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Young Subjects) | BI 409306 - 25 Milligram (mg) (Young Subjects) | BI 409306 - 50 Milligram (mg) (Young Subjects) | Placebo (Elderly Subjects) | BI 409306 - 25 Milligram (mg) (Elderly Subjects) | BI 409306 - 50 Milligram (mg) (Elderly Subjects) | Total
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 9 | 9 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] — As pre-specified in the protocol, the young and elderly subjects were analyzed separately. Population: Treated Set
  Years
    Young subjects: number analyzed (Participants) | 4 | 6 | 6 | 0 | 0 | 0 | 16
    Young subjects | 23.8 (3.0) | 34.7 (7.7) | 30.8 (10.2) |  |  |  | 30.5 (8.7)
    Elderly subjects: number analyzed (Participants) | 0 | 0 | 0 | 6 | 9 | 9 | 24
    Elderly subjects |  |  |  | 70.8 (3.4) | 69.9 (3.1) | 68.1 (2.4) | 69.5 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    Female | 3 | 1 | 2 | 2 | 5 | 4 | 17
    Male | 1 | 5 | 4 | 4 | 4 | 5 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was not reported in this trial Population: Treated Set
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 4 | 5 | 5 | 0 | 0 | 0 | 14
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
    White | 0 | 1 | 1 | 6 | 9 | 9 | 26
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Investigator Defined Drug-Related Adverse Events
Description: Percentage of subjects with investigator defined drug-related Adverse Events (AEs).
Time Frame: From the first administration of trial medication until 14 days after the last administration of trial medication, up to 28 days
Population: as for baseline characteristics
Measure: Number; unit: Percentage of subjects
Arm/Group | Placebo (Young Subjects) | BI 409306 - 25 Milligram (mg) (Young Subjects) | BI 409306 - 50 Milligram (mg) (Young Subjects) | Placebo (Elderly Subjects) | BI 409306 - 25 Milligram (mg) (Elderly Subjects) | BI 409306 - 50 Milligram (mg) (Elderly Subjects)
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 9 | 9
Percentage of subjects | 50.0 | 50.0 | 66.7 | 50.0 | 55.6 | 44.4

2. Secondary Outcome: Maximum Measured Concentration of the BI 409306 in Plasma (Cmax)
Description: Maximum measured concentration of the BI 409306 in plasma (Cmax).
Time Frame: PK blood samples were taken at 0, 0.167, 0.333, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 24 hours after drug administration.
Population: The pharmacokinetics (PK) set included all subjects in the treated set with at least 1 evaluable observation for a PK endpoint in at least 1 treatment period and no important protocol violations relevant to the PK evaluation. All subjects in the treated set who received active drug were included in the PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles per liter (nmol/L)
Arm/Group | BI 409306 - 25 Milligram (mg) (Young Subjects) | BI 409306 - 50 Milligram (mg) (Young Subjects) | BI 409306 - 25 Milligram (mg) (Elderly Subjects) | BI 409306 - 50 Milligram (mg) (Elderly Subjects)
Number analyzed (Participants) | 6 | 6 | 9 | 9
Nanomoles per liter (nmol/L) | 679 (44.1) | 1310 (33.9) | 459 (55.2) | 768 (55.3)

3. Secondary Outcome: Maximum Measured Concentration of the BI 409306 in Plasma at Steady State (Cmax, ss)
Description: Maximum measured concentration of the BI 409306 in plasma at steady state (Cmax, ss).
Time Frame: PK blood samples were taken at 312, 312.167, 312.333, 312.5, 312.75, 313, 313.5, 314, 314.5, 315, 316, 318, 320, 322, 324, 326, 336, 360, 384 hours after drug administration.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles per liter (nmol/L)
Arm/Group | BI 409306 - 25 Milligram (mg) (Young Subjects) | BI 409306 - 50 Milligram (mg) (Young Subjects) | BI 409306 - 25 Milligram (mg) (Elderly Subjects) | BI 409306 - 50 Milligram (mg) (Elderly Subjects)
Number analyzed (Participants) | 6 | 6 | 9 | 9
Nanomoles per liter (nmol/L) | 694 (33.1) | 1740 (29.8) | 516 (51.2) | 872 (56.3)

4. Secondary Outcome: Area Under the Concentration-time Curve of the BI 409306 in Plasma From 0 to 24 Hours (AUC0-24)
Description: Area under the concentration-time curve of the BI 409306 in plasma from 0 to 24 hours (AUC0-24).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles*hour per liter (nmol*h/L)
Arm/Group | BI 409306 - 25 Milligram (mg) (Young Subjects) | BI 409306 - 50 Milligram (mg) (Young Subjects) | BI 409306 - 25 Milligram (mg) (Elderly Subjects) | BI 409306 - 50 Milligram (mg) (Elderly Subjects)
Number analyzed (Participants) | 6 | 6 | 9 | 9
Nanomoles*hour per liter (nmol*h/L) | 1570 (33.5) | 2690 (50.2) | 622 (72.6) | 1030 (42.1)

5. Secondary Outcome: Area Under the Concentration-time Curve of the BI 409306 in Plasma at Steady State Over a Uniform Dosing Interval τ (AUCτ,ss)
Description: Area under the concentration-time curve of the BI 409306 in plasma at steady state over a uniform dosing interval τ (AUCτ,ss).
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles*hour per liter (nmol*h/L)
Arm/Group | BI 409306 - 25 Milligram (mg) (Young Subjects) | BI 409306 - 50 Milligram (mg) (Young Subjects) | BI 409306 - 25 Milligram (mg) (Elderly Subjects) | BI 409306 - 50 Milligram (mg) (Elderly Subjects)
Number analyzed (Participants) | 6 | 6 | 9 | 9
Nanomoles*hour per liter (nmol*h/L) | 1800 (29.7) | 3410 (40.8) | 682 (58.9) | 1250 (50.1)

6. Secondary Outcome: Time From Dosing to the Maximum Concentration of the BI 409306 in Plasma (Tmax)
Description: Time From Dosing to the Maximum Concentration of the BI 409306 in Plasma (tmax).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | BI 409306 - 25 Milligram (mg) (Young Subjects) | BI 409306 - 50 Milligram (mg) (Young Subjects) | BI 409306 - 25 Milligram (mg) (Elderly Subjects) | BI 409306 - 50 Milligram (mg) (Elderly Subjects)
Number analyzed (Participants) | 6 | 6 | 9 | 9
hours | 0.625 [0.333 to 1.500] | 0.750 [0.333 to 1.000] | 0.500 [0.333 to 0.750] | 0.500 [0.167 to 1.000]

7. Secondary Outcome: Time From Dosing to the Maximum Concentration of the BI 409306in Plasma at Steady State (Tmax,ss)
Description: Time From Dosing to the Maximum Concentration of the BI 409306in Plasma at Steady State (Tmax,ss).
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | BI 409306 - 25 Milligram (mg) (Young Subjects) | BI 409306 - 50 Milligram (mg) (Young Subjects) | BI 409306 - 25 Milligram (mg) (Elderly Subjects) | BI 409306 - 50 Milligram (mg) (Elderly Subjects)
Number analyzed (Participants) | 6 | 6 | 9 | 9
hours | 0.634 [0.500 to 1.500] | 0.417 [0.333 to 0.750] | 0.333 [0.333 to 0.550] | 0.367 [0.167 to 0.517]

8. Primary Outcome: Percentage of Subjects With Clinically Relevant Abnormalities for Different Tests
Description: Percentage of subjects with clinically relevant abnormalities in Vital signs,12-lead electrocardiogram (ECG), Clinical laboratory tests (hematology, clinical chemistry, and urinalysis), Physical examination, Suicidality assessment, Color discrimination test, Visual acuity test.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: Percentage of subjects with findings
Arm/Group | Placebo (Young Subjects) | BI 409306 - 25 Milligram (mg) (Young Subjects) | BI 409306 - 50 Milligram (mg) (Young Subjects) | Placebo (Elderly Subjects) | BI 409306 - 25 Milligram (mg) (Elderly Subjects) | BI 409306 - 50 Milligram (mg) (Elderly Subjects)
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 9 | 9
Percentage of subjects with findings
  Visual acuity test | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Color discrimination test | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Suicidality assessment | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Physical examination | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Clinical laboratory tests | 0.0 | 16.6 | 0.0 | 0.0 | 0.0 | 11.1
  12-lead electrocardiogram (ECG) | 25.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Blood pressure and pulse rate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Orthostatic intolerance | 25.0 | 0.0 | 0.0 | 33.3 | 33.3 | 0.0

ADVERSE EVENTS:
Time Frame: From the first administration of trial medication until 14 days after the last administration of trial medication, up to 28 days
Description: The treated set (TS) included all subjects who were randomised and documented to have taken at least one dose of investigational treatment.
Arm/Group | Placebo (Young Subjects) | Placebo (Elderly Subjects) | BI 409306 - 25 Milligram (mg) (Young Subjects) | BI 409306 - 50 Milligram (mg) (Young Subjects) | BI 409306 - 25 Milligram (mg) (Elderly Subjects) | BI 409306 - 50 Milligram (mg) (Elderly Subjects)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 2/4 | 3/6 | 3/6 | 4/6 | 6/9 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Young Subjects) (N=4) | Placebo (Elderly Subjects) (N=6) | BI 409306 - 25 Milligram (mg) (Young Subjects) (N=6) | BI 409306 - 50 Milligram (mg) (Young Subjects) (N=6) | BI 409306 - 25 Milligram (mg) (Elderly Subjects) (N=9) | BI 409306 - 50 Milligram (mg) (Elderly Subjects) (N=9)
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chromatopsia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 3
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eyelids pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 1 | 2 | 3 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 3 | 3 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3
Orthostatic intolerance (Nervous system disorders) | 1 | 2 | 0 | 0 | 3 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.